CLINICAL TRIAL: NCT00144495
Title: A Multicenter, Open-Label Study of Recombinant Human Erythropoietin in Anemic Cancer Patients Undergoing Chemotherapy
Brief Title: A Study of Recombinant Human Erythropoietin in Anemic Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPO308JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Chemotherapy Induced Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): patient whose ΔHb is less than 1.0g/dL on the day of 7th administration
  Interventions: Drug: recombinant human erythropoietin
- 2 (Experimental): patient whose ΔHb is 1.0g/dL or above on the day of 7th administration
  Interventions: Drug: recombinant human erythropoietin

INTERVENTIONS:
Drug: recombinant human erythropoietin — 3600IU(s.c.)/week for 7 weeks and 54000IU(s.c.)/week for 5 weeks
  Arms: 1
Drug: recombinant human erythropoietin — 36000IU(s.c.)/week for 12 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of recombinant human erythropoietin in anemic cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients

Exclusion Criteria:

* a history of myocardial, cerebral or pulmonary infarction
* severe hypertension beyond control by drugs

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2004-02; Primary Completion 2004-11 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The increase in Hb concentration | Day 28th or later

SECONDARY OUTCOMES:
Changes in QOL scores | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiharu Ishikura, Study Director — Chugai Pharmaceutical